CLINICAL TRIAL: NCT07383961
Title: LONG TERM FOLLOW UP AFTER PEDIATRIC SINGLE SITE ROBOTIC CHOLECYSTECTOMY
Status: Completed | Type: Observational
Sponsor: Good Samaritan Hospital Medical Center, New York (Other)
Responsible Party: Principal Investigator, Vinci Jones, Pediatric Surgeon, Good Samaritan Hospital Medical Center, New York
Other Study IDs: 25-005
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Robotic Surgical Procedure
Keywords: pediatric robotic surgery; single incision robotic surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic multiport cholecystectomy
- robotic single site cholecystectomy

SUMMARY:
Robotic single-site cholecystectomy (RSSC) was first reported in children the PI from GSH in 2015, demonstrating the feasibility, safety, and short learning curve associated with RSSC.

The primary advantages of RSSC identified in pediatric patients include superior cosmetic outcomes, reduced postoperative pain, and a shorter learning curve for surgeons compared to SILC. These benefits contribute to its growing acceptance among pediatric surgeons.

However, despite clear short-term benefits, the need for evaluating long-term outcomes in pediatric populations remains unmet. There are currently no studies reporting long-term complications or cosmetic satisfaction following RSSC in pediatric patients.

This study will attempt to evaluate the long term outcomes after RSSC and compare them with the current gold standard, multiport laparoscopic cholecystectomy, performed by the same surgeon at the same institution over a similar time frame.

DETAILED DESCRIPTION:
Robotic single-site cholecystectomy (RSSC) was first reported in children by Jones (2015), who conducted a retrospective review demonstrating the feasibility, safety, and short learning curve associated with RSSC compared to single-incision laparoscopic cholecystectomy (SILC) in pediatric patients, which has been proven to be technically challenging [1]. Subsequently, Esposito et al. further supported these findings, showing similar safety and effectiveness of RSSC in pediatrics over a 6-year period [2]. Rothenberg et al. compared robotic-assisted cholecystectomy (RC) to laparoscopic cholecystectomy (LC) in children, highlighting no significant differences in immediate postoperative complications, opioid utilization, or hospital readmissions but identifying higher costs associated with RC [3]. Kulaylat et al. similarly reported longer operative times (98 vs 79 minutes) and higher overall costs ($15,519 vs $11,197) for robotic procedures compared to laparoscopic ones, though postoperative complications and length of stay (LOS) were comparable [4].

The primary advantages of RSSC identified in pediatric patients include superior cosmetic outcomes, reduced postoperative pain, and a shorter learning curve for surgeons compared to SILC. These benefits contribute to its growing acceptance among pediatric surgeons.

However, despite clear short-term benefits, the need for evaluating long-term outcomes in pediatric populations remains unmet. There are currently no studies reporting long-term complications or cosmetic satisfaction following RSSC in pediatric patients.

In adult populations, short-term studies comparing RSSC and multiport laparoscopic cholecystectomy (MLC) revealed comparable hospital stay, complication rates, seroma formation, and infection rates [5]. Hagen et al. demonstrated increased costs and higher reoperation rates for hernias with RSSC compared to MLC in adults [6]. Lurje et al. evaluated short-term cosmetic outcomes, confirming patient satisfaction with robotic surgery in adults, but no pediatric data was provided [7].

In pediatric patients, short-term follow-ups primarily emphasized operative safety, operative time, hospital stay, and immediate postoperative complications, generally showing equivalence between RC and LC with the exception of higher costs for RC [3,4].

Long-term outcomes in adult populations show conflicting reports. Marks et al. demonstrated high patient-reported cosmetic satisfaction scores at 8-year follow-up favoring SILC over conventional laparoscopic surgery [8]. Conversely, Christoffersen et al. found that most incisional hernias following SILC occurred within two years post-surgery, suggesting the need for continued monitoring [9]. Recent adult cohort studies reported comparable operative times and hospital stays between robotic and laparoscopic procedures, but with slightly higher costs associated with robotic surgery [10].

The current literature underscores significant gaps in the long-term follow-up of pediatric RSSC outcomes. To date, comprehensive evaluation of long-term hernia rates, cosmetic satisfaction, and patient-reported outcomes in children undergoing RSSC is lacking. This study aims to fill this gap by providing essential long-term data on RSSC outcomes, affirming its durability and superiority as an alternative to MLC.

ELIGIBILITY:
Inclusion Criteria: Those who have undergone cholecystectomy by laparoscopic or robotic surgery over the past 12 years at GSUH -

Exclusion Criteria: multiple procedures at same time

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pediatric patients with gall bladder disease undergoing cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 24-60 months

SECONDARY OUTCOMES:
cosmetic satisfaction | 24-60months

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan University Hospital, West Islip, New York, United States

IPD SHARING:
Plan to Share IPD: No
IRB has limited patient information access only to the investigators